CLINICAL TRIAL: NCT06421688
Title: Effect of Vitamin C on Postoperative Pulmonary Complications After Intracranial: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Vitamin C on Postoperative Pulmonary Complications After Intracranial Tumor Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Dong Wang, Principal Investigator, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YXLL-KY-2024(039)
Record Dates: First submitted 2024-05-05; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Ascorbic Acid; Neurosurgical Procedures; Humans; Ventilator-Induced Lung Injury; Postoperative Complications
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Postoperative Complications | interventions — Ascorbic Acid; Sodium Chloride; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ascorbic acid group (Experimental): Patients received 50 mg/kg of Ascorbic acid after induction of anesthesia
  Interventions: Drug: Ascorbic acid
- Control comparator group (Placebo Comparator): Patients receive 50ml saline after induction of anesthesia
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ascorbic acid — After participants underwent induction of anesthesia, Ascorbic acid (Vitamin C Injection) was administered at a dosage of 50 mg/kg, diluted to 50 ml using saline, with a total amount not exceeding 4 g; pumping was performed using a micro pump at a rate of 25 ml/h.
  Other Names: vitamin C
  Arms: Ascorbic acid group
Drug: Saline — After participants underwent induction of anesthesia, 50 ml of saline was used and pumped using a micro pump at a rate of 25 ml/h.
  Other Names: saline (medicine)
  Arms: Control comparator group

SUMMARY:
The goal of this clinical trial is to investigate the effect of perioperative administration of vitamin C on postoperative pulmonary complications, with the aim of providing a safe and effective medication regimen for the prevention and treatment of postoperative pulmonary complications in patients undergoing surgery for craniocerebral tumors. The main questions it aims to answer are:

1. To determine whether vitamin C can reduce pulmonary complications after surgery for intracranial tumors.
2. Does intraoperative vitamin C improve the prognosis of surgical patients

Researchers will compare vitamin C to a placebo (saline) to see if vitamin C is effective for postoperative lung complications in patients undergoing surgery for cranial tumors.

1. Participants will be intravenously pumped with vitamin C for two hours after induction of anesthesia.
2. Participants will have intraoperative plasma sampling and recording of ventilator parameters, monitor parameters and perioperative data.
3. Participants will be followed up until discharge from the hospital to record symptoms and adverse events, and will be called at six months to check on their prognosis.

DETAILED DESCRIPTION:
Neurosurgery has a high incidence of postoperative pulmonary complications, increasing patient costs and affecting patient prognosis. Neurosurgery often requires hyperventilation to reduce intracranial pressure, so methods to reduce postoperative pulmonary complications such as small tidal volumes cannot be used routinely, and larger tidal volumes often result in injury to pulmonary endothelial cells, which leads to increased permeability of the pulmonary microvasculature, resulting in mechanically ventilated lung injury. Of course surgical injuries and mechanical ventilation can also cause oxidative stress injury to the lungs. Vitamin C is a common antioxidant drug and cofactor in the synthesis of many substances in the body, and many studies have shown that vitamin C prevents the increase in endothelial barrier permeability due to many causes. During the COVID-19 epidemic, vitamin C is seen as an important adjunct in preventing and ameliorating symptoms of COVID-19 patients. not only that, but vitamin C also assisted in postoperative analgesia and promote incision healing, so investigators would like to observe that by giving vitamin C during the surgery is able to prevent the occurrence of postoperative pulmonary complications or improve the prognosis of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need craniotomy treatment due to intracranial tumors;
2. age 18-75 years old;
3. American Society of Anesthesiologists classification: 1~3;
4. Patients and their families agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Patients with severe pulmonary infection or respiratory failure prior to surgery;
2. Patients with previous history of neurological or psychiatric diseases;
3. Patients with cardiac, hepatic and renal insufficiency;
4. patients who are receiving parenteral nutrition;
5. pregnant patients;
6. Patients ruled out by medication instructions;
7. Patients who require emergency surgery;
8. patients with combination of other malignant tumors;
9. patients who have participated in other clinical studies of drugs within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative pulmonary complications | About 10 days
  This will be assessed using the Postoperative Pulmonary Complications Score, which ranges from 0 to 5, with a score of ≥3 being considered positive for postoperative pulmonary complications. It was assessed every day before discharge and the highest score that occurred was recorded.

SECONDARY OUTCOMES:
Neuron-specific enolase levels | Post operative day 1
  Plasma levels of neuron-specific enolase, unit is ng/ml
Length of hospitalization | About 10 days
  Length of time between participant's completion of surgery and discharge
Oxygenation index | One hour postoperative
  PaO2/FiO2, in millimeters of mercury
Pain scores | 1 day, 3 days, 7 days postoperative
  Patient's postoperative pain level; Using a "Pain Visual Analogue Scale", a 10-centimeter-long ruler was used, with 0 indicating no pain and 10 representing the most intense pain that was intolerable. During the test, the participant points to the scale that best represents the level of pain, and the researcher assigns the participant a score based on the location of the point.
pulmonary compliance | Last hour of surgery.
  lung compliance in Milliliter/ centimeter water column
Interleukin-6 | 1 day, 3 days, 7 days postoperative
  The level of Interleukin-6 in the blood, in nanograms per liter
superoxide dismutase (SOD) | 1 day, 3 days, 7 days postoperative
  Blood levels of superoxide dismutase, in units per milliliter
body temperature | 1 day, 3 days, 7 days postoperative
  Postoperative body temperature in degrees Celsius
blood pressure | About 10 days
  Systolic and diastolic blood pressure，In millimeters of mercury
Brain-specific cardiolipin | About 3 days
  Plasma levels of brain-specific cardiolipin
neutrophil | About 10 days
  Levels of neutrophils in the blood, measured in units per liter.
C-reactive protein | 1 day, 3 days, 7 days postoperative
  Level of C-reactive protein in the blood in milligrams per liter

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wang, M.D, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data(IPD) will be available when this trial is finished and the article have been published

REFERENCES:
- [Background] Sogame LC, Vidotto MC, Jardim JR, Faresin SM. Incidence and risk factors for postoperative pulmonary complications in elective intracranial surgery. J Neurosurg. 2008 Aug;109(2):222-7. doi: 10.3171/JNS/2008/109/8/0222. PMID 18671633
- [Background] May JM, Harrison FE. Role of vitamin C in the function of the vascular endothelium. Antioxid Redox Signal. 2013 Dec 10;19(17):2068-83. doi: 10.1089/ars.2013.5205. Epub 2013 May 29. PMID 23581713
- [Background] Holford P, Carr AC, Jovic TH, Ali SR, Whitaker IS, Marik PE, Smith AD. Vitamin C-An Adjunctive Therapy for Respiratory Infection, Sepsis and COVID-19. Nutrients. 2020 Dec 7;12(12):3760. doi: 10.3390/nu12123760. PMID 33297491
- [Background] Wang D, Wang M, Zhang H, Zhu H, Zhang N, Liu J. Effect of Intravenous Injection of Vitamin C on Postoperative Pulmonary Complications in Patients Undergoing Cardiac Surgery: A Double-Blind, Randomized Trial. Drug Des Devel Ther. 2020 Aug 11;14:3263-3270. doi: 10.2147/DDDT.S254150. eCollection 2020. PMID 32848365
- [Background] Costa Leme A, Hajjar LA, Volpe MS, Fukushima JT, De Santis Santiago RR, Osawa EA, Pinheiro de Almeida J, Gerent AM, Franco RA, Zanetti Feltrim MI, Nozawa E, de Moraes Coimbra VR, de Moraes Ianotti R, Hashizume CS, Kalil Filho R, Auler JO Jr, Jatene FB, Gomes Galas FR, Amato MB. Effect of Intensive vs Moderate Alveolar Recruitment Strategies Added to Lung-Protective Ventilation on Postoperative Pulmonary Complications: A Randomized Clinical Trial. JAMA. 2017 Apr 11;317(14):1422-1432. doi: 10.1001/jama.2017.2297. PMID 28322416